CLINICAL TRIAL: NCT04750733
Title: Impact of Core Performance on Functional Parameters in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Feray Güngör, Physiotherapist, Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: 59491012-604.01.0
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; core stability; postural control; isokinetic strength; physical capacity; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis: Ambulatory MS patients
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Assessment of core strength and endurance, muscle strength, postural sway in different condition, physical capacity and fatigue

SUMMARY:
Optimal trunk control relies on somatosensory, motor and musculoskeletal integrity, which is often damaged in multiple sclerosis (MS). Researches on postural control in people with MS (PwMS) have revealed that reduced somatosensory conduction may adversely affect some functions. PwMS have increased postural sway in upright posture than healthy people. They move closer and slower when reaching out or taking a step. Trunk controls are weak and postural responses are delayed. The activation of core muscles is very important for an effective trunk control. Because the core region is considered a kinetic link that facilitates the transfer of torque and angular momentum between the upper and lower extremities during body movements. The decrease in core stability affects both trunk control and the quality of limb movements due to the kinetic chain in the body. There are a limited number of studies in the literature showing that core stability is reduced in PwMS. Our knowledge about the effects of this reduction on function in PwMS is very limited.

DETAILED DESCRIPTION:
The aim of this study is to evaluate core strength and endurance and determine its effect on postural control, knee muscle strength, physical capacity and fatigue parameters in individuals with MS. Also relationship between these parameters will investigate.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MS according to McDonald's criteria
* Disability level less than 6 according to EDSS (Expanded Disability Status Scale) score
* No attacks during the last 3 months
* Being an ambulatory
* Volunteering to participate in the study

Exclusion Criteria:

* Having orthopedic, neurological, psychological, etc. diseases that accompany MS and may affect treatment outcomes
* Doing regular sports
* Being involved in another physiotherapy and rehabilitation program related to MS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with MS followed in the Neurology Department of Bakirkoy Prof. Dr. Mazhar Osman Education and Research Hospital for Psychiatric and Neurological Diseases will be included.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Core strength | Baseline
  Core strength will be evaluated within the scope of core assessment. Curl-Up and Modified Push-Up test will be used for the evaluation of core strength.
Core endurance | Baseline
  Core endurance will be evaluated within the scope of core assessment. Trunk flexor, extensor, lateral endurance and plank will be used in the evaluation of core endurance and recorded as seconds.
Postural sway | Baseline
  Postural sways will be evaluated with biodex balance system in different condition such as open eyes on firm and foam surface, closed eyes on firm and foam surface, double stance on firm and foam surface, tandem stance on firm and foam surface.
İsokinetic strength | Baseline
  Concentric isokinetic muscle strength of the knee flexor and extensor muscles will be evaluated with Biodex isokinetic dynamometer at angular velocities of 30,60 and 90°/s.

SECONDARY OUTCOMES:
Physical capacity | Baseline
  Two-minute walk test (2-MWT) will be used to evaluate the mobility of the people with MS. 2-MWT is a measure of self-paced walking ability and functional capacity.
Mobility | Baseline
  Timed Up and Go (TUG) will be used. TUG is a test used to determine fall risk and measure the progress of balance, sit to stand and walking.
Fatigue | Baseline
  Fatigue Severity Scale (FSS) will be used to evaluate fatigue levels. This scale evaluates the severity of fatigue with 9 questions. Each question scores between 1 (I do not agree) and 7 (fully agree). The FSS score is the average value of nine sections. A high score indicates increased fatigue severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)